CLINICAL TRIAL: NCT03019133
Title: Prospective Randomized Controlled Trial to Compare and Analyze the Effects of Sound Masking and Reduction Techniques on Heart Rate and Blood Pressure Variability in Critically Ill Patients
Brief Title: Trial to Evaluate the Effects of Sound Modulation on Critically Ill Patients
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brian Gehlbach (Other)
Responsible Party: Sponsor-Investigator, Brian Gehlbach, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201609843
Record Dates: First submitted 2016-12-19; First posted 2017-01-12 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Physiological Stress; Delirium; Sleep Deprivation
Keywords: Heart rate; Blood pressure variability
MeSH Terms: conditions — Critical Illness; Delirium; Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (No Intervention): Usual care will be provided.
- Sound reduction (Active Comparator): Use of noise reduction headphones. Pro For Sho safety ear muffs with a noise reduction rate of 34dB will be used.
  Interventions: Device: Sound reduction
- Sound masking (Active Comparator): Use of headphones and relaxing music. Sennheiser HD 280 pro headphones will be used for sound masking.
  Interventions: Device: Sound masking

INTERVENTIONS:
Device: Sound reduction — Subjects will wear noise reduction headphones between the hours of 8:00 pm and 8:00 am.
  Arms: Sound reduction
Device: Sound masking — Subjects will wear wear headphones playing relaxing music between the hours of 8:00 pm and 8:00 am.
  Arms: Sound masking

SUMMARY:
The goal of the project is to determine the effects of noise masking and noise reduction on stress related physiological parameters in critically ill patients admitted to the intensive care unit.

DETAILED DESCRIPTION:
Sleep deprivation is common in critically ill patients in the intensive care unit (ICU) and may impair recovery. While noise is widely cited as the most common cause of sleep disruption in the ICU setting, its contribution to sympathetic activity in critically ill patients is not known. This is an important knowledge gap, because noise initiates a sequence of physiological changes including vasoconstriction, raised diastolic blood pressure, pupil dilatation and muscle tension. Furthermore, noise is implicated in sympathetic arousals, resulting in a release of adrenaline which prevents relaxation and consequently prevents the patient from falling asleep.

The investigators plan to study the effect of noise masking and noise reduction on stress related physiological parameters in critically ill patients admitted to the ICU. Subjects will be randomized into 3 separate groups: control, noise reduction, and noise masking. The investigators will compare the heart rate and blood pressure variability between and within the groups to determine the effects of treatment assignment on these variables. Non-invasive measurements obtained from the bedside monitor will be collected using physiological data acquisition software.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-99 years who are expected to receive care on an adult critical care unit for at least 24 hours

Exclusion Criteria:

* Admission for drug overdose or with a known substance abuse disorder
* Untreated sleep apnea disorder, narcolepsy, REM sleep behavior disorder, parasomnia, restless leg syndrome or other sleep disorder
* Use of hearing aids, or known significant conductive or sensory hearing loss
* Ventilator support via an endotracheal tube
* Use of vasopressors
* Unresponsive or delirious
* Subjects with known Dementia, Parkinson's disease, or other neurodegenerative disorder
* Subjects with a pacemaker or who have received cardiac transplant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Nocturnal LF/HF ratio (a.u.) | Day 1 of study
  The effect of group assignment on nocturnal (8pm to 8am) low frequency/high frequency (LF/HF) ratio will be determined.

SECONDARY OUTCOMES:
Nocturnal heart rate (bpm) | Day 1 of study
  The effect of group assignment on nocturnal (8pm to 8am) heart rate will be determined.
Nocturnal RMSSD (ms) | Day 1 of study
  The effect of group assignment on nocturnal (8pm to 8am) root mean square of sequential differences of RR intervals (RMSSD) will be determined.
Nocturnal blood pressure (mm Hg) | Day 1 of study
  The effect of group assignment on nocturnal (8pm to 8am) blood pressure (mean arterial pressure) will be determined.
Incidence of ICU delirium | Assessed at the time of ICU discharge up to a maximum of 28 days after enrollment, and averaging 4 days after enrollment
  The effect of group assignment on the incidence of ICU delirium as assessed by the CAM-ICU will be determined.
Hospital length of stay (days) | Assessed at the time of hospital discharge up to a maximum of 28 days after enrollment, and averaging 6 days after enrollment.
  The effect of group assignment on hospital length of stay will be assessed.
ICU length of stay (days) | Assessed at the time of ICU discharge up to a maximum of 28 days after enrollment, and averaging 4 days after enrollment.
  The effect of group assignment on ICU length of stay will be assessed.
Hospital mortality (%) | Assessed at the time of hospital discharge up to a maximum of 28 days after enrollment, and averaging 6 days after enrollment.
  The effect of group assignment on in-hospital mortality will be assessed.
Discharged home (%, versus discharge to another health care facility or died) | Assessed at the time of hospital discharge up to a maximum of 28 days after enrollment, and averaging 6 days after enrollment.
  The effect of group assignment on being discharged directly to home (versus to another skilled care facility or died) from the hospital will be assessed.

OTHER OUTCOMES:
Intra-individual nocturnal LF/HF ratio (a.u.) | Days 1 and 2 of study
  For each subject, the effect of treatment assignment on nocturnal (8pm to 8am) low frequency/high frequency (LF/HF) ratio will be determined by comparing the LF/HF ratio on Day 1 (intervention) with that on Day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Brian K Gehlbach, MD, Principal Investigator — Faculty
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, there are no definite plans for sharing individual participant data at this time.

REFERENCES:
- Available data/document: Informed Consent Form: 201609843 — http://hawkirb.research.uiowa.edu